CLINICAL TRIAL: NCT03133767
Title: Saline vs. Lactated Ringers for Emergency Department IV Fluid Resuscitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicholas M Mohr (Other)
Responsible Party: Sponsor-Investigator, Nicholas M Mohr, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201701764
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Fluid Loss; Symptom Complex, Triple; Emergencies
Keywords: Normal saline; Lactated ringers; Emergency department
MeSH Terms: conditions — Behcet Syndrome; Emergencies | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Fluid being administered to participants will be covered by an opaque bag. The investigator calling the participant for follow-up does not know how the participant was allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lactated ringers solution (Experimental): Participants in this arm will receive two liters of IV Lactated Ringer's solution during their emergency department stay
  Interventions: Drug: Lactated Ringer Solution
- Normal saline solution (Experimental): Participants in this arm will receive two liters of IV 0.9% sodium chloride solution during their emergency department stay
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag

INTERVENTIONS:
Drug: Lactated Ringer Solution — 2 liters of intravenous lactated ringers solution will be administered by peripheral IV
  Arms: Lactated ringers solution
Drug: Normal Saline 0.9% Infusion Solution Bag — 2 liters of intravenous normal saline solution will be administered by peripheral IV
  Arms: Normal saline solution

SUMMARY:
Administration of intravascular (IV) fluid is the most common emergency department (ED) procedure. IV fluids are integral to increasing effective blood volume and ensuring organ perfusion in patients with volume depletion and dehydration. There are many options of IV fluids providers can use when treating ED patients. Surveys show physicians do not cite an evidence-based reason for selecting the crystalloid IV fluid used; the decision was likely to be influenced by type and location of practice. A gap exists in the current literature, as there is no evidence for the optimal IV fluid choice for the ED patient requiring IV fluid before discharge.

Normal saline (NS) is commonly used as an IV fluid replacement in ED patients. However, NS has been associated with increased risk of acidosis and acute kidney injury. This study will use a novel approach of a patient-centered outcome in a non-critically ill population to ascertain the optimal IV fluid for patient quality of recovery. The results of this study will inform provider's IV fluid decisions between NS and LR. More importantly, the results of this study will have the power to improve patient's quality of recovery following IV fluid administration and subsequent ED discharge.

ED patients will be recruited, and participants will be randomized to receive one of two IV solutions (Lactated ringer's or normal saline). Participants will answer a survey before and after the intervention to assess their quality of recovery. The post-survey will be administered by phone after ED discharge. Participants will also be contacted by text message one week following their ED visit to gather information on their healthcare utilization.

DETAILED DESCRIPTION:
This is a single-center randomized, single-blinded, controlled clinical trial testing superiority of LR compared to NS in patients receiving IV fluid before discharge.

The study site is the University of Iowa Emergency Department (annual patient volume is 60,000 patients/year).

The study population will include adult ED patients presenting with chief complaints associated with volume depletion. Figure 1 outlines the enrollment flowchart for the study with inclusion and exclusion criteria. Research assistants (RAs) are available in the ED from 9am - 10pm every day, and an automated paging system will alert the team when patients qualify, as the study team has done previously. All participants will receive 2 liters of blinded IV fluid as part of the study. The intervention group will receive lactated ringer's, and the control group will receive normal saline (0.9% sodium chloride). Nursing staff will establish the peripheral IV access, and subjects will be blinded to group.

The primary outcome, Quality of Recovery-40, will be analyzed using a t-test (if parametric) or Mann Whitney U Test (non-parametric) in an intention-to-treat (ITT) analysis. Normality will be assessed with a Kolmogorov-Smirnov (K-S) and visualization of data. Due to the nature of time-critical emergency department research, an additional analysis will be done by treatment received and compared to the primary ITT analysis as a sensitivity analysis. Secondary outcomes will be reported as a relative risk with 95%CI in an ITT analysis. A safety analysis of secondary outcomes will be performed by treatment received (see page 37). Baseline characteristics will be reported with summary statistics as appropriate (mean, SD, median, IQR) and differences in characteristics will be conducted using a t-test and chi-square test, as appropriate. The following variables will also be assessed: actual fluid administered(mL), pre-intervention QoR-40 score, and time from intervention to primary outcome. If differences in these characteristics exist between the control and intervention groups, multivariate linear regression and multivariate logistic regression (primary and secondary outcomes, respectively) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient
* Chief complaint of nausea, vomiting or emesis, diarrhea, abdominal pain, dehydration, heat stroke or exhaustion
* ED provider approves administration of two liters of fluid
* ED provider states patient is likely to be discharged
* Patient has followed up with PCP in the last two years
* Patient has access to phone for next two days following ED discharge

Exclusion Criteria:

* Prisoners
* Children
* Women known to be pregnant
* Jaundice
* Current chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friederich A, Martin N, Swanson MB, Faine BA, Mohr NM. Normal Saline Solution and Lactated Ringer's Solution Have a Similar Effect on Quality of Recovery: A Randomized Controlled Trial. Ann Emerg Med. 2019 Feb;73(2):160-169. doi: 10.1016/j.annemergmed.2018.07.007. Epub 2018 Aug 23. PMID 30146446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
Started | 79 | 78
Completed | 41 | 53
Not Completed | 38 | 25
Not completed — Lost to Follow-up | 38 | 24
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactated Ringers Solution | Normal Saline Solution | Total
Number analyzed (Participants) | 41 | 53 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [22 to 41] | 39 [25 to 45] | 35 [23 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 24 | 58
  Male | 7 | 29 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 34 | 45 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 41 | 53 | 94

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery-40 Score at 24 Hours
Description: The Quality of Recovery-40 (QoR-40) is a validated instrument that quantifies patient's self-assessment of functional recovery, symptoms, and physical comfort. The QoR-40 scores range from 40 to 200 with a 200 representing a better recovery outcome. The survey consists of 40 questions scored from one to five with a Likert scale, and the total score is the sum of each question.
Time Frame: 24 hours after ED visit
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
Number analyzed (Participants) | 41 | 53
units on a scale | 166.8 [160.5 to 173.1] | 164.4 [157.8 to 171.0]
Statistical Analysis 1: Comparison: Lactated Ringers Solution vs Normal Saline Solution; Test type: Superiority; p = 0.608, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Quality of Recovery-40 Score After Administration
Description: as for outcome 1
Time Frame: Immediately after fluid administration
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
Number analyzed (Participants) | 41 | 53
units on a scale | 152.6 [145.3 to 159.9] | 141.6 [133.5 to 149.7]
Statistical Analysis 1: Comparison: Lactated Ringers Solution vs Normal Saline Solution; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants That Filled an ED Prescription
Description: Seven days after study enrollment, participants were asked by text message, "Have you filled any prescriptions from the emergency department?"
Time Frame: 7 days after study enrollment
Population: Only participants that received an ED prescription and responded to the seven-day text message were included in this analysis (26 participants in the LR and 25 in the NS group).
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
Number analyzed (Participants) | 26 | 25
Participants | 14 | 19
Statistical Analysis 1: Comparison: Lactated Ringers Solution vs Normal Saline Solution; Test type: Superiority; p = 0.202, Chi-squared

4. Secondary Outcome: Number of Participants That Returned to the ED Within 7 Days for the Same Complaint
Description: Seven days after study enrollment, participants were asked by text message, "Have you returned to the emergency department for the same problem?"
Time Frame: 7 days
Population: Response rates for the secondary outcomes were 47.4% (n=36) in the NS group and 53.3% (n=42) in the LR group.
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
Number analyzed (Participants) | 42 | 36
Participants | 5 | 7
Statistical Analysis 1: Comparison: Lactated Ringers Solution vs Normal Saline Solution; Test type: Superiority; p = 0.361, Chi-squared

5. Secondary Outcome: Participants That Sought Care From Another Healthcare Provider for the Same Complaint
Description: Seven days after study enrollment, participants were asked by text message, "Have you seen another medical provider for the same complaint?".
Time Frame: 7 days
Population: Response rates for the secondary outcomes were 47.4% (n=36) in the NS group and 53.3% (n=42) in the LR group.
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
Number analyzed (Participants) | 42 | 36
Participants | 9 | 7
Statistical Analysis 1: Comparison: Lactated Ringers Solution vs Normal Saline Solution; Test type: Superiority; p = 0.509, Chi-squared

ADVERSE EVENTS:
Time Frame: Participants could be assessed for adverse events at the phone call 24-48 hours following study enrollment and/or at the text message seven days following study enrollment.
Description: Participants responding to the 24-hour phone call and/or the seven-day text could be assessed for adverse events. Therefore, the total of participants in the LR group is 42 (one participant did not respond to the primary outcome, but did respond to the seven-day text to assess secondary outcomes).
Arm/Group | Lactated Ringers Solution | Normal Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/53
Other Adverse Events (participants affected / at risk) | 0/42 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03133767/Prot_SAP_000.pdf